CLINICAL TRIAL: NCT02055443
Title: Myocardial Ischemia Detection for Early Identification of Patients With Ischemic Chest Pain
Acronym: MID-EPIC
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Salah Shafiq Al-Zaiti, Assistant Professor of Acute & Tertiary Care, University of Pittsburgh
Other Study IDs: PRO13070234
Record Dates: First submitted 2014-01-30; First posted 2014-02-05 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Cardiac Ischemia; Chest Pain; Shortness of Breath
Keywords: nuclear cardiology; chest pain; cardiac ischemia; shortness of breath; ECG; EKG; electrocardiogram
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Holter monitor group: 12-lead holter monitor application
  Interventions: Other: 12-lead holter monitor application

INTERVENTIONS:
Other: 12-lead holter monitor application — -- The study coordinator will then obtain a 5-minute baseline high resolution (1000 samples/second), 12-lead resting ECG stream using H12+ holter ECG machine (Mortara Instruments, Milwaukee, WI). This ECG will be performed before the subject completed their clinical stress test.
  * The patient will then complete the scheduled nuclear stress test that involves exercise treadmill testing followed by single-photon emission computerized tomography (SPECT) scan as per hospital protocols. The exercise treadmill test and SPECT nuclear imaging scan are clinical in nature, and therefore, separate from the research study.
  * After completing the scheduled exam, the study coordinator will obtain another 5-minute 12-lead ECG stream prior to removing the chest electrodes but before their nuclear scan.
  Other Names: H12+ holter ECG machine (Mortara Instruments, Milwaukee, WI)

SUMMARY:
The purpose of this study is to evaluate whether new novel markers from the clinical electrocardiogram (EKG), which have been used as non-invasive measures of heart disease, can detect coronary artery disease in patients with chest pain. The researchers are especially interested in studying how changes in these unique waves evolve over time with rest and activity. It is hoped that the findings will be helpful in differentiating patients with cardiac chest pain at emergency departments from those with non-cardiac chest pain, as early identification can accelerate treatment and save lives.

Eligible participants are those age 18 and older who have been referred for a nuclear stress test at University of Pittsburgh Medical Center Presbyterian Hospital to rule out coronary artery disease as part of their clinical care.

DETAILED DESCRIPTION:
Acute Coronary Syndrome (ACS) is the leading cause of death worldwide. Differentiating ACS from other non-ischemic chest pain is imperative in emergency medicine and missed myocardial infarction remains one of the highest sources of medical malpractice in Emergency Departments (ED). At the same time, economic pressures and limited resources demand that physicians avoid hospital admission or protracted observation for every patient with chest pain or suspicious symptoms. In the absence of clear ST elevation (STE) on the electrocardiogram (ECG), ED providers have no reliable tools to quickly triage non-STE (NSTE) ACS patients. Current guidelines rely on blood biomarkers (e.g. cardiac enzymes) to identify this syndrome and do not completely describe ischemic ECG changes associated with it. ED Providers will need to delay the management of these high risk patients until cardiac biomarkers are withdrawn, analyzed, and interpreted. This results in greater mortality rates in NSTE-ACS patients and overburdens the healthcare system. The prolonged observation times at EDs and unnecessary admissions are just additional consequences that overuse nursing times and exacerbate nursing shortage.

ECG changes other than ST elevation and dynamic ECG changes are a rich opportunity for improving diagnostics. This proposal intends to provide new insights into how ischemic repolarization changes evolve over time in the subacute phase of myocardial ischemia. Sixty patients with suspected coronary artery disease referred for nuclear cardiac stress testing will be included. Resting 12-lead ECGs will be obtained before the stress test and one after the stress test but before the nuclear scan. Alterations in novel, computerized T wave indices will be correlated with focal myocardial ischemia seen on nuclear scans. Repeated Measures ANOVA with between group comparisons, and Generalized Estimation Equation will be used in the analysis. The results will provide insight on the diagnostic value of different novel T wave indices to detect myocardial ischemia. Results from this study will provide tools for ED providers to distinguish ACS from non-ischemic chest pain patients early in the triage process, especially in the absence of STE that constitutes the common standard nowadays.

ELIGIBILITY:
Inclusion Criteria:

* adults > 18 years of age
* referred for nuclear cardiac stress testing for suspected coronary artery disease.

There will be no restrictions to sex or race. Children and teens are less likely to have ischemic etiology of chest pain, justifying their exclusion. To optimize the clinical utility, there will be no exclusion criteria based on previous medical history, medications, or presenting chief complaint; all consecutive patients will be eligible.

Exclusion Criteria:

* Patients with un-interpretable ECGs or their ECG shows known secondary repolarization abnormalities (i.e. bundle branch blocks, ventricular hypertrophy, channelopathies, early repolarization) will be excluded. Of note, as per clinical guidelines, these patients do not get usually referred for exercise treadmill testing. This will improve the recruitment process of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Myocardial ischemia | 1-2 days per hospital SPECT protocol
  The primary outcome is the presence of radionuclide evidence of focal myocardial ischemia evidenced on nuclear cardiac stress testing (SPECT results).

CONTACTS AND LOCATIONS:
Overall Officials: Salah Shafiq Al-Zaiti, PhD, Principal Investigator — University of Pittsburgh School of Nursing
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States